CLINICAL TRIAL: NCT00004583
Title: A Randomized, Double-Blind, Phase III Study of ABT-378/Ritonavir Plus Stavudine and Lamivudine vs Nelfinavir Plus Stavudine and Lamivudine in Antiretroviral Naive HIV-Infected Subjects
Brief Title: A Phase III Study Comparing Two Different Anti-HIV Drug Combinations in HIV-Positive Patients Without Previous Anti-HIV Drug Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 285C; M98-863
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2009-02-20 (Estimated); Status verified 2009-02

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Administration, Oral; Stavudine; HIV Protease Inhibitors; Lamivudine; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Nelfinavir; ABT 378
MeSH Terms: conditions — HIV Infections | interventions — Lopinavir; Nelfinavir; Lamivudine; Stavudine

INTERVENTIONS:
Drug: Lopinavir/Ritonavir
Drug: Nelfinavir mesylate
Drug: Lamivudine
Drug: Stavudine

SUMMARY:
The purpose of this study is to see how safe a new protease inhibitor (PI) is and how well it fights HIV infection. A PI is a drug that stops HIV from using healthy cells to make more virus. This study will compare the new PI combination of ABT-378 plus ritonavir (RTV) with another PI, nelfinavir (NFV).

Earlier studies suggest ABT-378/RTV will be just as good as and perhaps better than NFV at fighting HIV infection.

DETAILED DESCRIPTION:
Based on the accumulated studies to date, it is expected that ABT-378/ritonavir will provide efficacy that is at least as good as (or superior to) nelfinavir when used in combination with reverse transcriptase inhibitors.

Patients are equally randomized to one of two treatment arms. In one arm, approximately 330 patients receive ABT-378/ritonavir plus nelfinavir placebo. In the other arm, approximately 330 patients receive nelfinavir plus ABT-378/ritonavir placebo. In both arms, these protease inhibitors are blinded to the investigator, patient, and sponsor. Both arms receive open-label stavudine and lamivudine. Vital sign measurements, physical examinations, ECGs, routine clinical laboratory evaluations, and determinations of antiviral and immunologic activity are performed at intervals throughout the study.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this trial if you:

* Are HIV positive.
* Have a viral load (level of HIV in your blood) of more than 400 copies/ml.
* Are age 12 or older.
* Agree to practice abstinence or use effective methods of birth control during the study.

Exclusion Criteria

You will not be eligible for this trial if you:

* Have taken anti-HIV drugs for more than 14 days in the past, or if you have ever taken d4T or 3TC.
* Are seriously ill or have an AIDS-related infection.
* Are pregnant or breast-feeding.
* Are taking certain medications.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 660
Dates: Start 1999-03

CONTACTS AND LOCATIONS:
Locations (83):
- United States (42):
  - Pacific Oaks Med Group, Beverly Hills, California
  - Orange County Ctr for Special Immunology, Fountain Valley, California
  - AIDS Healthcare Foundation, Los Angeles, California
  - Tower ID Med Associates, Los Angeles, California
  - UCLA CARE Ctr, Los Angeles, California
  - San Francisco Veterans Administration Med Ctr, San Francisco, California
  - Harbor - UCLA Med Ctr, Torrance, California
  - Yale Univ / AIDS Clinical Trials Unit, New Haven, Connecticut
  - Steinhart Medical Associates, Miami, Florida
  - Univ of Miami School of Medicine, Miami, Florida
  - Infectious Disease Research Institute, Tampa, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Emory Univ, Atlanta, Georgia
  - AIDS Research Alliance - Chicago, Chicago, Illinois
  - Division of Inf Diseases/ Indiana Univ Hosp, Indianapolis, Indiana
  - Univ of Kansas School of Medicine, Wichita, Kansas
  - Tulane Univ Med School, New Orleans, Louisiana
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Boston Med Ctr, Boston, Massachusetts
  - Community Research Initiative of New England, Brookline, Massachusetts
  - Univ of Michigan Hospitals and Health Ctrs, Ann Arbor, Michigan
  - Abbott Northwestern Hosp, Minneapolis, Minnesota
  - East Orange Veterans Administration Med Ctr, East Orange, New Jersey
  - Beth Israel Med Ctr, New York, New York
  - Cornell Clinical Trials Unit - Chelsea Clinic, New York, New York
  - Howard Grossman, New York, New York
  - SUNY at Stony Brook / Div of Infectious Disease, Stony Brook, New York
  - Duke Univ Med Ctr / Infectious Disease Clinic, Durham, North Carolina
  - Holmes Hosp / Univ of Cincinnati Med Ctr, Cincinnati, Ohio
  - Associates in Med and Mental Health, Tulsa, Oklahoma
  - Oregon Health Sciences Univ, Portland, Oregon
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - Stephen Hauptman, Philadelphia, Pennsylvania
  - The Miriam Hosp, Providence, Rhode Island
  - Vanderbilt Univ Med Ctr, Nashville, Tennessee
  - Central Texas Med Foundation, Austin, Texas
  - Oaklawn Physicians Group, Dallas, Texas
  - Univ of Texas Southwestern Med Ctr, Dallas, Texas
  - Joseph C Gathe, Houston, Texas
  - Infectious Disease Physicians Inc, Annandale, Virginia
  - Univ of Virginia Health Sciences Ctr, Charlottesville, Virginia
  - Univ of Wisconsin, Madison, Wisconsin
- Australia (3):
  - Royal Brisbane Hosp, Herston
  - Royal Perth Hosp, Perth
  - Alfred Hosp, Prahan
- Pulmologisches Zentrum Der Stadt Wien, Vienna, Austria
- Brazil (5):
  - Hosp Evandro Chagas Fioernz, Manguinhos RJ
  - Castelo, São Paulo
  - Fundacao Zerbini Casa Da Aids, São Paulo
  - Hosp Do Servidor Publico Estadual De Sao Paulo, São Paulo
  - Hosp Heliopolis, São Paulo
- Canada (6):
  - Saint Paul's Hosp, Vancouver, British Columbia
  - Ottawa General Hospital, Ottawa, Ontario
  - Toronto Gen Hosp, Toronto, Ontario
  - Clinique Medicale du Quartier Latin, Montreal, Quebec
  - Clinique Medicale L'Actuele, Montreal, Quebec
  - Montreal Chest Institute, Montreal, Quebec
- Denmark (2):
  - Righospitalet, Copenhagen
  - Hvidovre Univ Hosp, Hvidovre
- France (4):
  - Centre Hospitalier De Compiegne, Compiègne
  - CHU De Bicetre, Paris
  - Groupe Hospitalier Bichat-Claude Bernard, Paris
  - Hopital Paul Brousse, Villejuif
- Germany (5):
  - EPIMED, Berlin
  - Univ Zu Koeln, Cologne
  - Heinrich Heine Universitat, Düsseldorf
  - Klinikum Der Johann Wolfgang Goethe Universitat, Frankfurt
  - Allgemeines Krankenhaus St Georg, Hamburg
- Ctr of AIDS Diagnosis and Treatment, Warsaw, Poland
- Clinical Research Puerto Rico Inc, San Juan, Puerto Rico
- South Africa (3):
  - Miller, Belford Gardens
  - Cyrildene, Johannesburg
  - Wits Medical School, Parktown
- Spain (6):
  - Hosp Germans Trias I Pujol, Barcelona
  - Hosp Carlos III, Madrid
  - Hosp De Mostoles, Madrid
  - Hosp Doce De Octubre, Madrid
  - Hosp La Paz, Madrid
  - Hosp Virgen Del Rocio, Seville
- Universitatsspital Zurich, Zurich, Switzerland
- United Kingdom (3):
  - Brighton Gen Hosp, Brighton
  - Imperial College School of Medicine, London
  - Royal Free Hosp, London

REFERENCES:
- [Background] Murphy RL, Brun S, Hicks C, Eron JJ, Gulick R, King M, White AC Jr, Benson C, Thompson M, Kessler HA, Hammer S, Bertz R, Hsu A, Japour A, Sun E. ABT-378/ritonavir plus stavudine and lamivudine for the treatment of antiretroviral-naive adults with HIV-1 infection: 48-week results. AIDS. 2001 Jan 5;15(1):F1-9. doi: 10.1097/00002030-200101050-00002. PMID 11192874